CLINICAL TRIAL: NCT03868644
Title: HIV Prevention Among Youth: A Randomized Controlled Trial of Voluntary Counseling and Testing for HIV and Male Condom Distribution in Rural Kenya
Brief Title: The Impact of VCT and Condom Distribution as HIV Prevention Strategies Among Youth in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abdul Latif Jameel Poverty Action Lab (Other)
Collaborators: Innovations for Poverty Action (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0809002873R010
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: HIV/AIDS; HSV-2 Infection
Keywords: Youth; Kenya; Voluntary Counseling and Testing for HIV; Condoms; HIV prevention; HSV-2
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Seroconversion; Condoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Voluntary Counseling and Testing for HIV (VCT) (Experimental): Youth are offered VCT conducted onsite via mobile clinics in accordance with Kenya National HIV Testing Guidelines by certified VCT counselors trained by the National AIDS and STI Control Program (NASCOP).
  Interventions: Behavioral: Voluntary Counseling and Testing for HIV (VCT)
- Condoms (Experimental): Youth are offered 50 packages containing 3 condoms each of Trust brand condoms free of charge.
  Interventions: Behavioral: Condoms
- VCT and Condoms (Experimental): Youth are offered both VCT and condoms.
  Interventions: Behavioral: Voluntary Counseling and Testing for HIV (VCT); Behavioral: Condoms
- Control (No Intervention): No intervention is provided (beyond the standard available HIV prevention services within the area)

INTERVENTIONS:
Behavioral: Voluntary Counseling and Testing for HIV (VCT) — Youth are offered VCT conducted onsite via mobile clinics in accordance with Kenya National HIV Testing Guidelines by certified VCT counselors trained by the National AIDS and STI Control Program (NASCOP).
  Arms: VCT and Condoms; Voluntary Counseling and Testing for HIV (VCT)
Behavioral: Condoms — Youth are offered 50 packages containing 3 condoms each of Trust brand condoms free of charge.
  Arms: Condoms; VCT and Condoms

SUMMARY:
The vast majority of new HIV infections occur in sub-Saharan Africa, where nearly 2 million people become infected with HIV/AIDS every year. Forty-five percent of these new HIV infections occur among people under 25 years old, and nearly all of them are due to unprotected sex. Ensuring the adoption of safer sexual behavior among youth is critical to keeping the new generations free of HIV.

This research study aims to examine, through a large randomized controlled trial, the impact of two HIV prevention strategies among a youth population in Kenya: Voluntary Counseling and Testing for HIV (VCT), and condom distribution.

ELIGIBILITY:
Inclusion Criteria:

Youth previously participated in an earlier study by Duflo, Dupas and Kremer in 328 primary schools in the same study site in Western Province, Kenya who consent to participate.

Exclusion Criteria:

Youth sampled for the study who do not consent to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10646 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2014-07-01 (Actual)

PRIMARY OUTCOMES:
HSV-2 prevalence | 2 years post-intervention
  Assessed via a blood test

SECONDARY OUTCOMES:
% of youth who have high HIV knowledge | 2 years post-intervention
  Assessed via a questionnaire
% of youth who did not use a condom at last intercourse | 2 years post-intervention
  Assessed via a questionnaire
% of youth who reported having an STI or symptoms of an STI | 2 years post-intervention
  Assessed via a questionnaire
% of youth who report ever being pregnant | 2 years post-intervention
  Assessed via a questionnaire
Number of sexual partners | 2 years post-intervention
  Assessed via a questionnaire
HIV prevalence | 2 years post-intervention
  Assessed via a blood test
% of youth who have accepting attitudes towards people living with HIV (PLHIV) | 2 years post-intervention
  Assessed via a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Esther Duflo, Principal Investigator — Massachusetts Institute of Technology; Pascaline Dupas, Principal Investigator — Stanford University; Vandana Sharma, Principal Investigator — Harvard School of Public Health (HSPH)

REFERENCES:
- [Derived] Duflo E, Dupas P, Ginn T, Barasa GM, Baraza M, Pouliquen V, Sharma V. HIV prevention among youth: A randomized controlled trial of voluntary counseling and testing for HIV and male condom distribution in rural Kenya. PLoS One. 2019 Jul 30;14(7):e0219535. doi: 10.1371/journal.pone.0219535. eCollection 2019. PMID 31361767